CLINICAL TRIAL: NCT00859339
Title: A Phase II Trial of Neoadjuvant Cisplatin, Gemcitabine and Sunitinib Malate Followed by Radical Cystectomy for Transitional Cell Carcinoma (TCC) of the Bladder: Hoosier Oncology Group GU07-123
Brief Title: Neoadjuvant Cisplatin, Gemcitabine, Sunitinib Malate + Radical Cystectomy for TCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient Toxicities
Sponsor: Noah Hahn, M.D. (Other)
Collaborators: Pfizer (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Noah Hahn, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG GU07-123
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Transitional Cell Carcinoma of the Bladder
Keywords: TCC
MeSH Terms: interventions — Gemcitabine; Cisplatin; Sunitinib; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Treatment (Experimental): Neoadjuvant cisplatin, gemcitabine and sunitinib malate followed by radical cystectomy
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Sunitinib Malate; Procedure: Radical Cystectomy

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine ( 1000 mg/m2) IV days 1 and 8
Drug: Cisplatin — Cisplatin (70 mg/m2) IV day 1
Drug: Sunitinib Malate — Sunitinib malate (37.5 mg) oral daily for days 1-14
Procedure: Radical Cystectomy — Radical cystectomy performed no sooner than 2 weeks but within 6 weeks of the last dose of sunitinib malate.

SUMMARY:
This trial will investigate the activity of sunitinib combined with cisplatin and gemcitabine followed by radical cystectomy in patients with Transitional Cell Carcinoma (TCC) of the Bladder.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Gemcitabine ( 1000 mg/m2) IV days 1 and 8
* Cisplatin (70 mg/m2) IV day 1 and
* Sunitinib malate (37.5 mg) oral daily for days 1-14

The treatment regimen will be administered in four, 21-day, cycles followed by radical cystectomy performed no sooner than 2 weeks but within 6 weeks of the last dose of sunitinib malate.

ECOG performance status 0 or 1

Hematopoietic:

* Absolute Neutrophil Count (ANC) > 1.5 K/mm3 [(IS): 1.5 x 109/L]
* Platelets > 100 K/mm3 [(IS): 100 x 109/L]
* Hemoglobin (Hgb) > 9.0 g/dL [(IS): 90 g/L]

Hepatic:

* Total bilirubin < 1.5 x Upper Limit of Normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN

Renal:

* Calculated creatinine clearance of > 60 cc/min

Cardiovascular:

* No uncontrolled angina, congestive heart failure or myocardial infarction or coronary/peripheral artery bypass graft within 6 months prior to registration for protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of muscle-invasive transitional cell carcinoma of the bladder (stage II-III) with no evidence of metastatic disease (focal squamous and/or adenocarcinoma differentiation allowed, sarcomatoid and small-cell components not allowed). Patient with any degree of fixation of the pelvic sidewall are not eligible.
* Must be willing to undergo a cystoscopy if tumor block is not available prior to registration for protocol therapy.
* Eligible for radical cystectomy as per the attending urologist.
* Prior radiation therapy to bone marrow is allowed to < 25% of the marrow, and must be completed at least 6 months prior to registration for protocol therapy
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years at the time of consent.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.

Exclusion Criteria:

* No prior radiotherapy to the pelvis.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason< grade 7 prostate cancers, or other cancer for which the patient has been disease-free for at least 5 years.
* No treatment with any investigational agent within 30 days prior to registration for protocol therapy.
* No cerebrovascular accident or transient ischemic attack within 6 months prior to registration for protocol therapy.
* No evidence of pulmonary embolism within 6 months prior to registration for protocol therapy.
* No uncontrolled hypertension (>150/100 mm Hg despite optimal medical therapy).
* No evidence of ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade 2.
* No history of uncontrolled/untreated thyroid dysfunction.
* No prolonged QTc interval (> 450 msec) on pre-entry electrocardiogram obtained within 28 days prior to being registered on study.
* Patients on warfarin (>2mg) for thrombosis must be able and willing to switch to low molecular weight heparin prior to registration for protocol therapy.
* No use of drugs having proarrhythmic potential (terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide and flecainide) within 7 days prior to registration for protocol therapy.
* No use of CYP3A4 inhibitors (see section 5.3 for a list) within 7 days of registration for protocol therapy.
* No use of CYP3A4 inducers (see section 5.3 for a list) within 14 days of registration for protocol therapy.
* No use of amiodarone (CYP3A4 inhibitor) within 6 months of registration for protocol therapy.
* Females must not be breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Hahn, M.D., Study Chair — Hoosier Cancer Research Network
Locations (5):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Baylor College of Medicine, Houston, Texas
- St. Bartholomew's Hospital (Barts), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galsky MD, Hahn NM, Powles T, Hellerstedt BA, Lerner SP, Gardner TA, Yu M, O'Rourke M, Vogelzang NJ, Kocs D, McKenney SA, Melnyk AM Jr, Hutson TE, Rauch M, Wang Y, Asmar L, Sonpavde G. Gemcitabine, Cisplatin, and sunitinib for metastatic urothelial carcinoma and as preoperative therapy for muscle-invasive bladder cancer. Clin Genitourin Cancer. 2013 Jun;11(2):175-81. doi: 10.1016/j.clgc.2012.10.001. Epub 2012 Dec 8. PMID 23228446
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- CGS + Radical Cystectomy: Neoadjuvant cisplatin, gemcitabine and sunitinib malate followed by radical cystectomy
  Gemcitabine: Gemcitabine ( 1000 mg/m2) IV days 1 and 8
  Cisplatin: Cisplatin (70 mg/m2) IV day 1
  Sunitinib Malate: Sunitinib malate (37.5 mg) oral daily for days 1-14
  Radical Cystectomy: Radical cystectomy performed no sooner than 2 weeks but within 6 weeks of the last dose of sunitinib malate.
Period: Overall Study
Arm/Group | CGS + Radical Cystectomy
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CGS + Radical Cystectomy
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 70 [48 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 7
  United Kingdom | 2

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate.
Description: number of participants with a pCR
Time Frame: 18 months
Population: 8 participants were evaluable for pCR
Measure: Number; unit: particpants with pCR
Arm/Group | CGS + Radical Cystectomy
Number analyzed (Participants) | 8
particpants with pCR | 2

2. Secondary Outcome: Safety Profile
Description: Evaluate the safety profile of Neoadjuvant Cisplatin, Gemcitabine, Sunitinib Malate + Radical Cystectomy in participants with TCC
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | CGS + Radical Cystectomy
Number analyzed (Participants) | 9
participants
  Perioperative bleeding | 4
  neutropenia | 2
  neutropenic fever | 1
  thrombocytopenia | 1
  anemia | 1
  nausea/emesis | 3
  syncope | 2
  myocardial infarction | 1
  fatigue | 1

3. Secondary Outcome: Objective Response Rate
Description: To determine the objective response rate for patients with measurable disease according to RECIST.
Time Frame: 18 months
Population: No data was collected or analyzed for the secondary objective due to termination of the trial (toxicity)
Arm/Group | CGS + Radical Cystectomy
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival
Time Frame: 18 months
Population: No data was collected or analyzed for the secondary objective due to termination of the trial (toxicity)
Arm/Group | CGS + Radical Cystectomy
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlate Biomarker Expression
Description: To evaluate the impact of sunitinib malate in combination with cisplatin and gemcitabine on expression of selected biomarkers.
Time Frame: 18 months
Population: No data was collected or analyzed for the secondary objective due to termination of the trial (toxicity)
Arm/Group | CGS + Radical Cystectomy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From on-study to off-study, a maximum of four cycles plus time for recovery and radical cystectomy, a maximum of six months.
Arm/Group | CGS + Radical Cystectomy
Serious Adverse Events (participants affected / at risk) | 7/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGS + Radical Cystectomy (N=9)
CARDIAC ISCHEMIA/INFARCTION (Cardiac disorders) | 1 (1)
HEMORRHAGE, GU / BLADDER (Gastrointestinal disorders) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / KIDNEY (Infections and infestations) | 1 (1)
INFECTION - OTHER (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / WOUND (Infections and infestations) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
OBSTRUCTION, GU / BLADDER (Renal and urinary disorders) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 1 (1)
ULCER, GI / ESOPHAGUS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGS + Radical Cystectomy (N=9)
ANOREXIA (Gastrointestinal disorders) | 2 (2)
BLADDER SPASMS (Renal and urinary disorders) | 1 (1)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 2 (4)
CREATININE (Investigations) | 4 (6)
DEHYDRATION (Gastrointestinal disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 3 (3)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
EDEMA: LIMB (Blood and lymphatic system disorders) | 3 (3)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 6 (10)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 1 (2)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 2 (2)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 1 (2)
HEMOGLOBIN (Blood and lymphatic system disorders) | 5 (13)
HEMORRHAGE, GU / BLADDER (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE/BLEEDING ASSOCIATED WITH SURGERY, INTRA-OPERATIVE OR POSTOPERATIVE (Injury, poisoning and procedural complications) | 4 (4)
HYPERTENSION (Cardiac disorders) | 2 (2)
HYPOTENSION (Cardiac disorders) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BLADDER (URINARY) (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 3 (3)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 3 (8)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (5)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTRAOCULAR (Eye disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (3)
NEUROPATHY: SENSORY (Nervous system disorders) | 1 (1)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 5 (11)
OBSTRUCTION, GU / BLADDER (Renal and urinary disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 2 (2)
PAIN / BLADDER (Renal and urinary disorders) | 2 (2)
PAIN / BUTTOCK (General disorders) | 1 (1)
PAIN / CARDIAC/HEART (Cardiac disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / HEAD/HEADACHE (General disorders) | 1 (1)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN - OTHER (General disorders) | 1 (2)
PLATELETS (Blood and lymphatic system disorders) | 3 (6)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 2 (3)
THYROID FUNCTION, LOW (HYPOTHYROIDISM) (Endocrine disorders) | 1 (2)
URINE COLOR CHANGE (Renal and urinary disorders) | 1 (2)
VOMITING (Gastrointestinal disorders) | 2 (3)
WEIGHT LOSS (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to pre-defined stopping rules (patient toxicities)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No